CLINICAL TRIAL: NCT04936113
Title: An Open-Label, Multicenter Study to Evaluate Continued Safety of FB-401 for up to 48 Weeks in Children, Adolescent and Adult Subjects (Ages 2 Years and Older) With Mild to Moderate Atopic Dermatitis Previously Enrolled in FB401-01 Phase 2 Study
Brief Title: Continued Safety Evaluation of FB-401 in Children, Adolescents and Adults (2 Years and Older) With Mild to Moderate Atopic Dermatitis Previously Enrolled in the FB401-01 Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure of the Phase 2 study (protocol FB401-01) to meet its endpoint.
Sponsor: Forte Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FB401-02
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; microbiome; probiotic; commensal Gram-negative bacteria; transdermal water loss; allergic diseases; dermatitis; eczema; skin diseases; skin diseases, eczematous; immune system diseases
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema; Skin Diseases; Skin Diseases, Eczematous; Immune System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FB-401 (Experimental): FB-401 applied topically
  Interventions: Biological: FB-401

INTERVENTIONS:
Biological: FB-401 — Topical

SUMMARY:
The purpose of this study is to evaluate the continued safety and tolerability of FB-401 in subjects 2 years of age or older with mild to moderate atopic dermatitis. FB-401 will be applied topically for up to 48 additional weeks and subjects will be evaluated for safety.

ELIGIBILITY:
Inclusion Criteria:

* Participated in Protocol FB401-01, completed through Week 20 visit and able to directly enroll into this (FB401-02) study
* Refrain from use of all other atopic dermatitis treatments, unless given permission by medical monitor

Exclusion Criteria:

* Subject experienced a serious adverse event or severe adverse event attributable to study drug in Protocol FB401-01
* Severe concomitant illness that, in the Investigator's opinion, would adversely affect subject participation in the study, whether medical or psychological
* Pregnant (or planning to become pregnant during the period of the study) or lactating females

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 52 weeks
  Safety evaluations

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - MedaPhase, Inc, Newnan, Georgia
  - DS Research, Clarksville, Indiana
  - DS Research, Louisville, Kentucky
  - Cyn3rgy Research, New Brighton, Minnesota
  - Cyn3rgy Research, Gresham, Oregon
  - Bellaire Dermatology Associates, Bellaire, Texas

REFERENCES:
- [Background] Myles IA, Earland NJ, Anderson ED, Moore IN, Kieh MD, Williams KW, Saleem A, Fontecilla NM, Welch PA, Darnell DA, Barnhart LA, Sun AA, Uzel G, Datta SK. First-in-human topical microbiome transplantation with Roseomonas mucosa for atopic dermatitis. JCI Insight. 2018 May 3;3(9):e120608. doi: 10.1172/jci.insight.120608. PMID 29720571